CLINICAL TRIAL: NCT01639404
Title: Allogeneic Umbilical Cord Blood Therapy for Children With Cerebral Palsy
Brief Title: Umbilical Cord Blood Therapy for Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MinYoung Kim, M.D. (Other)
Responsible Party: Sponsor-Investigator, MinYoung Kim, M.D., Associate Professor, Bundang CHA Hospital
Organization: Bundang CHA Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPUCB
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Umbilical Cord Blood; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Umbilical Cord Blood and Rehabilitation (Experimental): Allogeneic Umbilical Cord Blood Administration and Active Rehabilitation
  Interventions: Procedure: Umbilical Cord Blood Administration; Other: Active Rehabilitation

INTERVENTIONS:
Procedure: Umbilical Cord Blood Administration — The subjects will be undertaken allogeneic umbilical cord blood infusion intravenously or intraarterially under non-myeloablative immunosuppression.
  Other Names: Donated Umbilical Cord Blood Units from Affiliated Cord Blood Bank
Other: Active Rehabilitation — All subjects should participate in active rehabilitation. They will receive two physical and occupational therapy sessions per day. Post discharge, each participant should continue to receive rehabilitation therapy at least 3 days per week until the study completion.

SUMMARY:
This study aims to evaluate the efficacy of umbilical cord blood therapy for children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy is a disorder of movement and posture resulted from a non-progressive lesion or injury of the immature brain. It is a leading cause of childhood onset disability.

Many experimental animal studies have revealed that umbilical cord blood is useful to repair neurological injury in brain.

On the basis of many experimental studies, umbilical cord blood is suggested as a potential therapy for cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy with abnormal muscle tone
* Gross Motor Function Classification System (GMFCS): I, II, III, IV, V
* Willing to comply with all study procedure

Exclusion Criteria:

* Medical illnesses including pneumonia or renal function at enrollment
* Presence of known genetic disease
* Presence of drug hypersensitivity which is related to this study remedy
* Poor cooperation of guardian,including inactive attitude for rehabilitation and visits for follow-up
* Decision by the principal investigator when there are unexpected events that may affect the outcomes

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Changes in Motor Performance | Baseline - 1 month - 3 months
  GMPM (Gross Motor Performance Measure) as a standardized measurement tool for assessing quality of movement regarding 3 properties of 5 ones; alignment, coordination, dissociated movement, stability, and weight shift (range: 0~100, Higher value means better motor quality). GMPM scores at each assessment time points will be reported.
Changes in Standardized Gross Motor Function | Baseline - 1 month - 3 months
  GMFM (Gross Motor Function Measure) as a standardized measurement tool for assessing Gross Motor Function consisting of sub-scales; lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping (range: 0~100 , Higher value means better gross motor function). GMFM scores at each assessment time points will be reported.

SECONDARY OUTCOMES:
Changes in Cognitive Neurodevelopmental Outcome | Baseline - 1 month - 3 months
  Korean version of Bayley Scale of Infant Development-II (K-BSID-II) Mental Scales (higher value means better mental function: 0 - worst, 178 - best). K-BSID-II Mental Scale raw scores at each assessment time points will be reported.
Changes in Motor Neurodevelopmental Outcome | Baseline - 1 month - 3 months
  Korean version of Bayley Scale of Infant Development-II (K-BSID-II) Motor Scales (higher value means better motor function: 0 - worst, 112 - best). K-BSID-II Motor Scale raw scores at each assessment time points will be reported.
Changes in Functional Independence in Daily Activities | Baseline - 1 month - 3 months
  WeeFIM (Functional Independence Measure for Children) measures functional independence in daily activities. WeeFIM contains 18 items and each item is ranked from complete dependence (scored as 1) to complete independence (scored as 7). The range is from 18 to 126 and higher scores mean more independent performance in daily activities. Total WeeFIM scores measured at each assessment time points will be reported.
Changes in Visual Perception Test | Baseline - 1 month - 3 months
  Visual perception function will be evaluated with one of three measures: DTVP (Developmental Test of Visual Perception), MVPT (Motor-free Visual Perception Test), and VMI (Visual-Motor Integration, Visual Perception and Motor Coordination). All can be scored as percentile rank from 0 to 100. Higher values mean better visual perception ability.
Changes in Muscle Strength | Baseline - 1 month - 3 months
  Summation of MMT (manual muscle strength test score): summated scores of the manual muscle strength test (zero=0, trace=1, poor=2, fair=3, good=4, normal=5) for flexors, extensors, abductors, and adductors of bilateral shoulder and hip joints; flexors and extensors of bilateral elbow, wrist, and knee; dorsiflexors and plantar flexors of the ankles (range: 0 ~ 160) Higher scores mean better muscle strength. Categories of outcome table will be summation of MMT scores measured at each assessment time point.
Changes in Functional Performance in Daily Activities | Baseline - 1 month - 3 months
  Pediatric Evaluation of Disability Inventory (PEDI) for assessing functional performance in daily activities in children (All values are adjusted and higher value means better functional performance, 0 - worst, 100 - best). We will report 2 scales and 3 domains of each scale: a Functional Skill Scale (FSS) and a Caregiver Assistance Scale (CAS) which are divided respectively into 3 domains: self care, mobility, and social function. Categories of outcome table will be each domain scores measured at each assessment time point.

CONTACTS AND LOCATIONS:
Overall Officials: MinYoung Kim, M.D., Ph.D., Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea